CLINICAL TRIAL: NCT00693290
Title: Improving Outcomes for Patients Requiring Oral Bowel Preparation for Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ulster (Other)
Collaborators: Action Cancer (Other); Western Health and Social Care Trust (Other)
Responsible Party: Mrs Daphne Garrett, Western Health & Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 07/NIR03/40
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Colorectal Cancer
Keywords: Colonoscopy; Colorectal screening; Colon preparation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sodium phosphate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Fleet plus low residue diet sheet.
  Interventions: Other: low residue diet
- 2 (No Intervention): No intervention, usual care, Fleet plus liquid only diet

INTERVENTIONS:
Other: low residue diet — Fleet (usual preparation) plus diet sheet for low residue diet
  Other Names: Sodium Phosphate
  Arms: 1

SUMMARY:
Study hypothesis The overall aim of this study is to compare two bowel preparations that are used prior to a colonoscopy procedure.

The principal research questions are:

1. Does the use of a low residue diet increase patient concordance to the bowel preparation instructions?
2. Does the use of a low residue diet decrease the adequacy of assessment of the mucosa?
3. Does the use of a low residue diet increase the willingness of patients to undertake repeated examination as is required for disease follow-up?
4. Does body weight affect perceived tolerability of either group?

ELIGIBILITY:
Inclusion Criteria:

* Patients attending for Colonoscopy.
* Patients referred for colonoscopy via General Practitioner.

Exclusion Criteria:

* Individuals who would not fully understand trial purpose (assessed by a cognisance scale if required)
* Previous episodes of total or partial small bowel obstruction
* Previous colonic surgery
* Known swallowing disorder
* Pregnancy
* Extremes of age (Less than 16 or greater than 80)
* Small Intestine disorders
* Renal Insufficiency (Serum Creatinine> 110)
* Congestive Heart failure
* Presence of ascites
* Severe Colitis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Clarity of the mucosa evaluated by the Ottawa Scale. | At endoscopy screening

SECONDARY OUTCOMES:
Concordance with the bowel preparation. | Prior to the endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Garrett, Principal Investigator — Western Health and Social Care Trust
Locations (1):
- Western Health and Social Care Trust, Londonderry, Northern Ireland, United Kingdom